CLINICAL TRIAL: NCT06590207
Title: Administering Convalescent Plasma Rich With Neutralizing Abs. to Hospitalized Adults With WNV - a Double-blind Randomized Controlled Study
Brief Title: Convalescent Plasma for the Treatment of Patients With WNV - a Double- Blind Randomized Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Gili Regev-Yochay MD, Infection Prevention & Control Unit, Director, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1381-24-SMC
Record Dates: First submitted 2024-07-31; First posted 2024-09-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-07

CONDITIONS: West Nile Fever With Neurologic Manifestation (Diagnosis); West Nile Fever Without Complications
Keywords: WNV; Neutralizing Abs; Convalescent plasma; neuroinvasive
MeSH Terms: conditions — Disease | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be conducted in a double-blind manner - the preparation/placebo will be provided by the pharmacy in a sealed bag.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 200ml of neutralizing plasma (Experimental): The plasma of the convalescents: produced in the blood bank of Sheba Medical Center, from the blood of Sheba workers who participated in the SPRI study (Helsinki 0196-23) and whose blood was found to have neutralizing antibodies to WNV (above 1:524). The blood units from the volunteers who will donate will meet all the requirements of a normal blood donation and will only include men or women who were not pregnant, and the units will pass all the tests accepted at the blood bank before donation.
  Interventions: Drug: plasma rich with WNV neutralizing antibodies
- Saline (Placebo Comparator): 200 ml Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: plasma rich with WNV neutralizing antibodies — 200 ml plasma of the convalescents: produced in the blood bank, from the blood of Sheba workers who participated in the SPRI study (Helsinki 0196-23) and whose blood was found to have neutralizing antibodies to WNV above 1:524. The blood units from the volunteers who will donate will meet all the requirements of a normal blood donation and will only include men or women who were not pregnant, and the units will pass all the tests accepted at the blood bank before donation.
  Other Names: Neurtalizing plasma
  Arms: 200ml of neutralizing plasma
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
Name of the study:

Administering neutralizing convalescent plasma to hospitalized patients with West Nile fever - a double-blind randomized controlled study.

The purpose of this study is to test the safety and effectiveness of giving blood plasma from convalescents rich in neutralizers as treatment against West Nile fever.

DETAILED DESCRIPTION:
The study is performed in Sheba Medical Center ( and will be expanded in the soon future to other Medical centers in Israel).

Hospitalized patients diagnosed by blood/CSF PCR or IgM, with West Nile Virus will be recruited to the study.

After signing an informed consent they will be randomized (2:1) to receive either blood plasma rich in neutralizing antibodies or saline as placebo.

Number of participants in this center: 130 Age range: 60 years old and older, 18-60 years old with immunosuppression.

Inclusion criteria:

* Hospitalized patients with positive WNV-PCR with fever/neurological symptoms, and 72 hours have not yet passed since the positive result.
* Age 60 or older.
* Age over 18 and younger than 60 with immunosuppression (hypogammaglobulinemia, solid organ transplants, bone marrow transplants, hemato-oncological malignancies).

Exclusion criteria:

* Age younger than 60 without immunosuppression.
* More than 72 hours have passed since the diagnosis of West Nile fever.
* Pregnant women.

Reference to the inclusion of pregnant women, special populations - children and those lacking judgment- not relevant: excludes pregnant women and special populations.

The duration of the medical trial includes the follow-up period after the trial:

The duration of the treatment is one day, single dose of plasma/saline. The follow-up period is 90 days.

The clinical follow-up plan (during and at the end of the treatment):

A total of 10 visits will be conducted. On day 1, the following will be performed: screening, Medical history & Physical examination, IV Convalescent Plasma vs. Saline, Urine and blood for PCR, functional & neurologic assesment, IgG and IgM from serum, blood test for CBC & renal function.

On day 2-7 and 30 and 90, AE will be collected. On day 3, 5, 7 Urine and blood for PCR will be collected. Neurologic assesment will be conducted on all visits. Serology will be collected also on day 30 and 90.

After discharge, a follow-up visit will be performed either by a visit to the clinic or via phone call.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with positive WNV-PCR with fever/neurological symptoms, and 72 hours have not yet passed since the positive result.
* Age 60 or older.
* Age over 18 and younger than 60 with immunosuppression (hypogammaglobulinemia, solid organ transplants, bone marrow transplants, hemato-oncological malignancies).

Exclusion Criteria:

* Age younger than 60 without immunosuppression.
* More than 72 hours have passed since the diagnosis of West Nile fever.
* Pregnant women. Criteria for exclusion from the experiment: none Reference to the inclusion of pregnant women, special populations - children and those lacking judgment- not relevant: excludes pregnant women and special populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Unfavorable outcom = Composite outcome of mortality or functional deterioration on day 30 | day 28-32
  functional deterioration will be defined using Barthel Index

SECONDARY OUTCOMES:
unfavorable outcome on day 90 | day 88-92
  same as primary outcome but on day 90
Serious adverse events | day 2-32
  Allergic reaction, pulmonary congestion, hemolysis
Mortality | day 28-92
  Mortality by day 90
Functional deterioration by day 30 & 90 | 28-92 days
  decrease in Barthel index from pre-infection baseline
Neurologic deterioration by day 30 & 90 | 28-92 days
  combined neurologic score of Barthel index, glasgow outcome score and modified minimental score

OTHER OUTCOMES:
Mechanical ventilation | 2-92 days
  Mechanical ventilation
ICU | 2-92days
  ICU

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Va Smilovici-Ofir, Phd, Study Chair — Sheba research grants and academic collaboration director
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassal R, Shohat T, Kaufman Z, Mannasse B, Shinar E, Amichay D, Barak M, Ben-Dor A, Bar Haim A, Cohen D, Mendelson E, Lustig Y. The seroprevalence of West Nile Virus in Israel: A nationwide cross sectional study. PLoS One. 2017 Jun 16;12(6):e0179774. doi: 10.1371/journal.pone.0179774. eCollection 2017. PMID 28622360
- [Background] Planitzer CB, Modrof J, Kreil TR. West Nile virus neutralization by US plasma-derived immunoglobulin products. J Infect Dis. 2007 Aug 1;196(3):435-40. doi: 10.1086/519392. Epub 2007 Jun 18. PMID 17597458
- [Background] Srivastava R, Ramakrishna C, Cantin E. Anti-inflammatory activity of intravenous immunoglobulins protects against West Nile virus encephalitis. J Gen Virol. 2015 Jun;96(Pt 6):1347-1357. doi: 10.1099/vir.0.000079. Epub 2015 Feb 9. PMID 25667322
- [Background] Gnann JW Jr, Agrawal A, Hart J, Buitrago M, Carson P, Hanfelt-Goade D, Tyler K, Spotkov J, Freifeld A, Moore T, Reyno J, Masur H, Jester P, Dale I, Li Y, Aban I, Lakeman FD, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Lack of Efficacy of High-Titered Immunoglobulin in Patients with West Nile Virus Central Nervous System Disease. Emerg Infect Dis. 2019 Nov;25(11):2064-2073. doi: 10.3201/eid2511.190537. PMID 31625835
- [Background] Mbonde AA, Gritsch D, Harahsheh EY, Kasule SN, Hasan S, Parsons AM, Zhang N, Butterfield R, Shiue H, Norville KA, Reynolds JL, Vikram HR, Chong B, Grill MF. Neuroinvasive West Nile Virus Infection in Immunosuppressed and Immunocompetent Adults. JAMA Netw Open. 2024 Mar 4;7(3):e244294. doi: 10.1001/jamanetworkopen.2024.4294. PMID 38546642
- See also: Treatment and Prevention of West Nile Virus Disease — https://www.cdc.gov/west-nile-virus/hcp/treatment-prevention/index.html#:~:text=There%20is%20no%20specific%20treatment,of%20blood%20and%20organ%20donors.